CLINICAL TRIAL: NCT05706233
Title: Effect of Postoperative Erector Spinae Plane Block as a Rescue Pain Therapy in Patients Undergoing Laparoscopic Cholecystectomy: A Historical Cohort Study
Brief Title: Erector Spinae Plane Block as a Rescue Pain Therapy in Patients Undergoing Laparoscopic Cholecystectomy
Status: Completed | Type: Observational
Sponsor: Istanbul Saglik Bilimleri University (Other)
Responsible Party: Principal Investigator, Taner Abdullah, Specialist, Istanbul Saglik Bilimleri University
Other Study IDs: 2021.11.254
Record Dates: First submitted 2023-01-09; First posted 2023-01-31 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Regional Anesthesia Morbidity; Cholecystitis, Chronic
MeSH Terms: conditions — Cholecystitis; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Erector Spina Plane Block (ESPB)
  Interventions: Procedure: Erector Spina Plane Group
- Intravenous Group (IV)
  Interventions: Procedure: IV analgesic intervention

INTERVENTIONS:
Procedure: Erector Spina Plane Group — ESPB had been applied postoperatively: from T8 level, 20mL bupivacaine %0,5 + 5ml %2 lidocaine was applied.
  Groups: Erector Spina Plane Block (ESPB)
Procedure: IV analgesic intervention — IV analgesics had been applied: All meperidine boluses are dosed in line with the pain intensity as follows: 10 mg if NRS > 3, 20 mg if NRS > 5, 30 mg if NRS > 8. If NRS score is not reduced at least 20% when compared to prior one, additional meperidine bolus is applied.
  Groups: Intravenous Group (IV)

SUMMARY:
Laparoscopic cholecystectomy, one of the most commonly performed abdominal surgeries, is a gold standard therapy for surgical treatment of benign biliary diseases.

Erector spinae plane block (ESPB) was first presented in 2016 as the treatment of neuropathic pain in a case series, and gained popularity very quickly due to its safety applicability, and effect on both the visceral and parietal component of pain by providing paravertebral, transforaminal and epidural spread. Preoperative application of ESPB has taken its place as a part of multimodal analgesia in laparoscopic cholecystectomy cases over time and has been shown to reduce postoperative pain scores and opioid consumption and to improve quality of recovery scores. However, there is no data regarding the use of ESPB in the postoperative period as a rescue therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing laparoscopic cholecystectomy
* Patients with NRS>3 scores in the PACU

Exclusion Criteria:

* ASA > 2
* Violation of standart protocol (anesthesia and analgesia)
* application of ESPB preoperatively
* age > 65
* Surgery duration >90min or <45min

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients undergoing laparoscopic cholecystectomy
Sampling Method: Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2022-05-15 (Actual); Study Completion 2022-05-15 (Actual)

PRIMARY OUTCOMES:
effect of ESPB applied postoperatively on the meperidine consumption in PACU | 1 HOUR
  As part of the standardized perioperative care management, the pain intensity is evaluated with the numeric pain rating scale (NRS). If the NRS is > 3 meperidine bolus or ESPB is applied in line with the patients' selection and the patients are evaluated in every 5 min in terms of their NRS scores until NRS < 4 is achieved. If NRS score is not reduced at least 20% when compared to prior one, additional meperidine bolus is applied. All meperidine boluses are dosed in line with the pain intensity as follows: 10 mg if NRS > 3, 20 mg if NRS > 5, 30 mg if NRS > 8. NRS scores and meperidine boluses applied are recorded on the PACU follow-up form.

SECONDARY OUTCOMES:
effect of ESPB applied postoperatively on numeric rating scores in PACU | 1 HOUR
  As part of the standardized perioperative care management, the pain intensity is evaluated with the numeric pain rating scale (NRS). If the NRS is > 3 meperidine bolus or ESPB is applied in line with the patients' selection and the patients are evaluated in every 5 min in terms of their NRS scores until NRS < 4 is achieved. If NRS score is not reduced at least 20% when compared to prior one, additional meperidine bolus is applied. All meperidine boluses are dosed in line with the pain intensity as follows: 10 mg if NRS > 3, 20 mg if NRS > 5, 30 mg if NRS > 8. NRS scores and meperidine boluses applied are recorded on the PACU follow-up form.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Basaksehir Cam and Sakura City Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes